CLINICAL TRIAL: NCT06858358
Title: Comparison of Robotic-Assisted Medial Congruent and Conventional Medial Pivot Total Knee Arthroplasty: a Prospective, Multicenter Analysis
Brief Title: Robotic Medial Congruent Vs. Conventional Medial Pivot TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures (Other)
Collaborators: Iuliu Hatieganu University of Medicine and Pharmacy (Other); County Clinical Emergency Hospital Cluj-Napoca (Other)
Responsible Party: Principal Investigator, Marian Andrei Melinte, Principal investigator, George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rosa_MP_MC_3002025
Record Dates: First submitted 2025-02-21; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthristis
Keywords: Robotic; Knee arthroplasty; TKA; ROSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ROSA Robotic-assisted TKA with Zimmer Biomet Persona Medial Congruent implant (Experimental)
  Interventions: Procedure: Robotic assisted total knee arthroplasty
- Conventional TKA with Microport Evolution Medial-Pivot (Experimental)
  Interventions: Procedure: Conventional total knee arthroplasty (cTKA)

INTERVENTIONS:
Procedure: Robotic assisted total knee arthroplasty — • ROSA RATKA with Zimmer Biomet Persona Medial Congruent
  Arms: ROSA Robotic-assisted TKA with Zimmer Biomet Persona Medial Congruent implant
Procedure: Conventional total knee arthroplasty (cTKA) — cTKA with Microport Evolution Medial-Pivot
  Arms: Conventional TKA with Microport Evolution Medial-Pivot

SUMMARY:
This multicenter, prospective cohort study will evaluate whether Robotic-Assisted total knee arthroplasty (RATKA) with a Medial Congruent implant is a successful method to improve implant alignment, insert thickness accuracy, and patient satisfaction, compared to a conventional TKA (cTKA) Medial Pivot technique. It aims to assess and compare clinical and functional outcomes in patients with severe knee osteoarthritis at 3, 6, and 12 months.

DETAILED DESCRIPTION:
This prospective, non-randomized, multicenter trial evaluates robotic-assisted (ROSA® Robotic Platform with Zimmer Biomet Persona® Medial Congruent) versus conventional (MicroPort Evolution® Medial-Pivot) total knee arthroplasty (TKA) in approximately 300 adults with severe osteoarthritis. By comparing robotic precision with a well-established Medial-Pivot design, this investigation aims to clarify whether robotic-assisted TKA confers superior implant positioning, reduced alignment outliers, and enhanced patient-reported outcomes (PROMS). The primary outcome measures include insert thickness, alignment accuracy (outliers defined as >2° from the mechanical axis on full-leg radiographs), and patient satisfaction at 6 and 12 months. Two surgeons will perform both techniques, and one surgeon will perform only the conventional procedure. The 18-month study is conducted under local Institutional Review Board approvals (Medlife, Medicover, SCJU Cluj Napoca, Monza Bucuresti) and complies with GDPR. Results are intended for publication in a high-impact orthopedic journal. No external funding is provided.

ELIGIBILITY:
Inclusion Criteria:

Patients with severe osteoarthritis (greater than III Ahlback)

Exclusion Criteria:

Patients who refuse participation in the study Low-grade osteoarthritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Polyethylene insert thickness | Perioperative/ Periprocedural
  Insert Thickness: Measured and analyzed in millimeters
Mechanical axis outliers | Perioperative/ Periprocedural
  Outliers: Defined as more than 2.0 degrees from mechanical alignment, measured on full-leg X-ray

SECONDARY OUTCOMES:
International knee documentation committe (IKDC) subjective score | 3, 6, and 12 months post-operative
  The IKDC is a purely subjective assessment that assigns patients a functional overall rating. Three (3) categories are examined by the questionnaire: symptoms, athletic activity, and knee function. The symptoms subscale aids in evaluating issues like pain, stiffness, edema, and knee giving way.
  The ICC, which varies from 0.87 to 0.98, was deemed sufficient (>0.70). Overall, it was discovered that the IKDC-SKF has positive test-retest reliability (Grevnerts et al. 2015). The IKDC subjective form scored acceptable for construct validity (84% confirmation of the predefined hypotheses) and responsiveness (86% confirmation of the predefined hypotheses) (van Meer et al. 2015).
Forgotten joint score-12 (FJS-12) | 3, 6, and 12 months post-operative
  The primary objective of the FJS-12 is to evaluate the extent to which patients "forget" their artificial joints during daily activities. A higher score indicates that the patient is less aware of their joint, suggesting better surgical outcomes and higher levels of patient satisfaction.

CONTACTS AND LOCATIONS:
Locations (2):
- Romania (2):
  - MedLife Humanitas Hospital, Cluj-Napoca, Cluj
  - Medicover Cluj Hospital, Cluj-Napoca, Cluj